CLINICAL TRIAL: NCT05031039
Title: Skeletal and Dental Maturational Stages in a Sample of Egyptian Subjects With Cleft Lip and Palate Deformity: A Cross-Sectional Study
Brief Title: Skeletal and Dental Maturational Stages in a Sample of Egyptian Subjects With Cleft Lip and Palate Deformity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, omima khaled salah, orthodontist, master student, Cairo University
Other Study IDs: 14422018441165
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cleft Lip and Palate
Keywords: skeletal & dental maturational stages
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female Egyptian subjects with Cleft Lip and Palate Deformity: Egyptians females that have unilateral or bilateral cleft lip and palate deformity
- Male Egyptian subjects with Cleft Lip and Palate Deformity: Egyptians males that have unilateral or bilateral cleft lip and palate deformity

SUMMARY:
The aim of this research is to evaluate the skeletal and dental maturation of cleft lip and palate patients in a sample of Egyptian population using the CVM as indicator for the skeletal maturation and the Demirjian method as indicator for the dental one when compared to a group of Egyptian non-CLP subjects of the same age.

DETAILED DESCRIPTION:
Chronological age (CA) is not considered an accurate method for assessing the stage of physical or growth development of an individual in childhood or adolescence. For that reason, skeletal and dental maturation can be used in order to examine the rate of physical maturation of the population. Cervical vertebral maturation (CVM) method uses lateral cephalometric radiography to evaluate skeletal maturity. It is considered the preferable method due to its advantage of avoiding unnecessary extra radiation. The CVM method developed by Baccetti et al. (2005) depends on the morphology of the three cervical vertebrae (C2, C3, and C4), which divided skeletal growth into six stages of based on the morphology of the previously mentioned cervical vertebrae. The Demirjian method is considered as one of the most worldwide used method for assessment of the dental maturation due to its reliability. It depends on panoramic x-rays through which the dental developmental stage of 7 lower left teeth appears, and according to the gender of the patient the sum of values of the teeth will be transform to age through the standard tables of Carmen M. Nolla; 1960.

ELIGIBILITY:
Inclusion Criteria:

(1) Subjects with non-syndromic CLP aged 6-18 years. (2) Subjects with no CLP deformity, aged 6-18 years. (4) Patients having complete records comprising dental/medical history and a lateral cephalometric and panoramic radiograph.

(5) No congenitally missing teeth in the mandible. (6) No previous history of trauma to the face, neck.

Exclusion Criteria:

* Radiographs of poor quality.
* Any growth or hereditary or systematic diseases or syndromes
* Any trauma or fracture of the jaw that might have affected the normal growth of permanent dentition.

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Egyptian subjects with Cleft Lip and Palate Deformity
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
dental age | 5 months
  Dental age will be evaluated by the Demirjian method

SECONDARY OUTCOMES:
skeletal age | 5 months
  skeletal age will be measured using the cervical vertebral method that was modified by Baccetti 2005